CLINICAL TRIAL: NCT04968249
Title: Michigan eArly Disease Progression Cohort in COPD (MAP COPD)
Brief Title: Michigan Early Disease Progression Cohort
Acronym: MAP_COPD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, MeiLan Han, Professor, University of Michigan
Other Study IDs: HUM00176147
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: COPD
Keywords: Early COPD; COPD; Smoking; CAPTURE; RETHINC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and nasal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Gold 0: Participant must be ages 30-55 years; and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC ≥ 0.70 and FEV1 ≥ 80% predicted.
  Interventions: Other: Observational
- Gold 1: Participants shall be between ages 30-55 years, and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC < 0.70 and FEV1 >= 80% predicted.
  Interventions: Other: Observational
- Gold 2: Participants shall be between ages 30-55 years, and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC < 0.70 and FEV1 50-79% predicted.
  Interventions: Other: Observational
- Preserved Ratio Impaired Spirometry (PRISm): Participant shall be between ages 30-55 years and have: ≥10 year smoking history, post-bronchodilator of FEV1 50-79% predicted and a predicted FEV1/FVC ≥ 0.70.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational Cohort to understand risk factors for early COPD.

SUMMARY:
The aim of this project is to develop a disease progression cohort within the University of Michigan Health System to capture pulmonary function, symptom assessments and quantitative imaging among patients at risk for or with an established diagnosis of COPD, focusing however on "early" COPD (age 30-55 and GOLD stage 0,1, 2, and prism).

DETAILED DESCRIPTION:
Participants between the ages of 30-55 with at least 10 pack-year smoking history will be enrolled into a observational longitudinal cohort.

During the course of the study, additional funding was secured, so data could be collected for a 3-year period from participants. Some of the cohort are co-enrolled in another study (NCT05033990) where they received a CT scan as part of the study. Those participants will not be re-scanned during the course of this study.

ELIGIBILITY:
Inclusion Criteria:

* GOLD 0 Participant must be ages 30-55 years; and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC ≥ 0.70 and FEV1 ≥ 80% predicted.
* Preserved Ratio Impaired Spirometry (PRISm) participants shall be between ages 30-55 years; and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV150-79% predicted and FEV1/FVC > 0.70.
* GOLD 1 participants shall be between ages 30-55 years, and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC < 0.70 and FEV1 >= 80% predicted. OR
* GOLD 2 participants shall be between ages 30-55 years, and have: ≥ 10 pack-year smoking history; post-bronchodilator FEV1/FVC < 0.70 and FEV1 50-79% predicted.

Exclusion Criteria:

* Severe asthma, which is defined as any of the following:

Current (i.e., at the time of the visit) GINA Step 4 or higher therapy (medium dose ICS/LABA or high dose ICS or add-on LAMA; Medium dose = >250 fluticasone propionate =100 fluticasone furoate, >200 beclomethasone, >400 budesonide, >220 mometasone). We will accept low-dose ICS/LABA or medium dose ICS.

or 3 or more unscheduled healthcare visits (provider/urgent care/ER) for asthma in the past 12 months or One asthma hospitalization in the past 12 months

* Concurrent participation in a therapeutic trial where treatment is blinded.
* Active pregnancy at the time of the baseline or return visits. This special population is being excluded to minimize potential for fetal radiation exposure.
* Cognitive dysfunction that prevents the participant from completing study procedures.
* BMI > 35.0 kg/m2 at baseline, due to the effects of body weight on CT scan imaging quality.
* The presence of a respiratory condition other than COPD or asthma, or of a comorbid condition that in the judgment of the investigator may be the principal cause of respiratory symptoms (e.g., dyspnea or decreased exercise tolerance).
* Any illness expected to cause mortality in the next 3 years.
* Any implanted metallic devices or prosthesis above the waist that could degrade thoracic CT scan image quality.
* History of thoracic radiation or thoracic surgery with resection of lung tissue

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients meeting inclusion criteria who have established disease as well as smokers meeting inclusion criteria where pulmonary function testing has not been performed.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
CAAT score ≥ 10 | 3 years
  Proportion of individuals with CAAT score ≥ 10
Exacerbations in the prior year | 3 years
  Frequency of moderate and severe exacerbations in the prior year measured at baseline

SECONDARY OUTCOMES:
Radiographic abnormalities on baseline CT | 3 years
  Proportion of individuals with radiographic abnormality on baseline CT defined as PRMfSAD≥15% and/or PRMEmph ≥3%

CONTACTS AND LOCATIONS:
Overall Officials: MeiLan Han, Principal Investigator — University of Michigan, Michigan Medicine
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez FJ, Han MK, Allinson JP, Barr RG, Boucher RC, Calverley PMA, Celli BR, Christenson SA, Crystal RG, Fageras M, Freeman CM, Groenke L, Hoffman EA, Kesimer M, Kostikas K, Paine R 3rd, Rafii S, Rennard SI, Segal LN, Shaykhiev R, Stevenson C, Tal-Singer R, Vestbo J, Woodruff PG, Curtis JL, Wedzicha JA. At the Root: Defining and Halting Progression of Early Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Jun 15;197(12):1540-1551. doi: 10.1164/rccm.201710-2028PP. No abstract available. PMID 29406779